CLINICAL TRIAL: NCT07072208
Title: A Prospective and Exploratory Clinical Study of Pomalidomide, Rituximab and Orelabrutinib Combined With Polatuzumab Vedotin in the Treatment of Newly Diagnosed Elderly Patients With DLBCL
Brief Title: Pomalidomide, Rituximab and Orelabrutinib Combined With Polatuzumab Vedotin in the Treatment of Newly Diagnosed Elderly Patients With DLBCL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024471
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Polatuzumab vedotin; pomalidomide; rituximab; Diffuse Large B-Cell Lymphoma; elderly patients; orelabrutinib
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pro-pola regimen (Experimental): The study will start with an initial 21-days of induction therapy with Pro regimen (Pomalidomide, rituximab and orelabrutinib)，following imaging examinations to evaluate response rates. Patients not achieving mRR (defined as complete remission [CR], partial remission [PR], and mini response [miniR; lesion reduction: 25.0%-50.0%]) were withdrawn from the study. Patients achieving mRR (with a lesion reduction of ≥25%) received Pro-pola(Pro regimen plus polatuzumab vedotin), in a 21-day cycle for 6 cycles.
  Interventions: Drug: Induction therapy-Pro regimen; Drug: Consolidation therapy-Pro-pola regimen

INTERVENTIONS:
Drug: Induction therapy-Pro regimen — Pro regimen induction(21days per cycle*1 cycle)
  * Pomalidomide 4mg per tablet 4mg orally from Days 1 to 7 of each cycle
  * Rituximab 100mg per vial 375mg/m2, intravenous drip, Day 1 of each cycle
  * Orelabrutinib 50mg per tablet 150mg orally per day from Days 1 to 21 of each cycle
Drug: Consolidation therapy-Pro-pola regimen — Pro-pola regimen consolidation(21days per cycle*6 cycle) -Pomalidomide 4mg per tablet 4mg orally from Days 1 to 7 of each cycle -Rituximab 100mg per vial 375mg/m2, intravenous drip, Day 1 of each cycle -Orelabrutinib 50mg per tablet 150mg orally per day from Days 1 to 21 of each cycle -Polatuzumab vedotin 30mg per vial 1.8 mg/kg, intravenous drip, Day 1 of each cycle

SUMMARY:
To evaluate the efficacy and safety of the Pro-Pola （Pomalidomide, rituximab, orelabrutinib and polatuzumab vedotin) regimen in elderly patients (aged ≥70 years) with newly diagnosed diffuse large B-cell lymphoma (DLBCL).

DETAILED DESCRIPTION:
The study will start with an initial 21-days of induction therapy with Pro regimen (Pomalidomide, rituximab and orelabrutinib)，following imaging examinations to evaluate response rates. Patients with a lesion reduction of ≥25% received Pro-pola(Pro regimen plus polatuzumab vedotin), in a 21-day cycle for 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥70 years unfit or frail
2. There is at least one image-measurable lesion with a measurable lesion of at least 15 mm.
3. Histologically confirmed treatment-naive DLBCL.
4. Life expectancy is>3 months.
5. appropriate organ function: Cardiac function: Cardiac ejection fraction ≥50%; Liver function: alanine aminotransferase and aspartate aminotransferase ≤3 times the upper limit of normal; Renal function: Serum creatinine clearance ≥30mL/min; Lung function: SPO2 >90% without oxygen inhalation
6. Adequate bone marrow reserve is defined as:

   Hemoglobin ≥8g/dL, platelet count ≥75×10^9/L, Absolute neutrophil value ≥1.0×10^9/L, If accompanied by bone marrow invasion, platelet count ≥50×10^9/L, absolute neutrophil count ≥0.75×10^9/L.
7. Patients have the ability to understand and are willing to provide written informed consent.
8. Subjects with childbearing or childbearing potential must be willing to practice birth control from the date of registration in this study to the follow-up period of the study.

Exclusion Criteria:

1. Severe abnormal liver and kidney function (alanine aminotransferase, bilirubin, creatinine>3 times the upper limit of normal);
2. Presence of organic heart disease or severe arrhythmia leading to clinical symptoms or abnormal cardiac function (NYHA Functional Class Grade ≥2);
3. Uncontrolled active infection;
4. Co-existence of other tumors requiring treatment or intervention;
5. DLBCL involving central nervous system;
6. Current or expected need for systemic corticosteroid treatment;
7. Previous or current history of vascular embolism;
8. Other psychological conditions that prevent the patient from participating in the study or signing informed consent.
9. In the investigator's judgment, it is unlikely that the subject will complete all protocol-required study visits or procedures, including follow-up visits, or will not meet the requirements for participation in the study.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Complete response rate(CRR) | At the end of 6 cycles of Pro-pola regimen (each cycle is 21 days)
  The rate of patients who achieved CR after 6 cycles of Pro-pola regimen

SECONDARY OUTCOMES:
Objective response rate(ORR) | At the end of 6 cycles of Pro-pola regimen (each cycle is 21 days)
  The rate of patients who achieved CR or PR after 6 cycles of Pro-pola regimen
2-year progression-free survival(PFS) | From the enrollment to 2-year after the treatment of last patient
  PFS will be assessed from the start of the treament to date of progression, relapse, death or end of follow-up.
2-year overall survival(OS) | From the enrollment to 2-year after the treatment of last patient
  OS will be assessed from the start the treatment to date of death or end of follow-up.
Main adverse reactions | From the enrollment to 1 months after 6 cycles of Pro-pola regimen of the last patient (each cycle is 21 days)
  The safety of the therapeutic regimen measured by the major adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Zhengming Jin, Study Chair — The First Affiliated Hospital of Soochow University; Changju Qu, Study Director — The First Affiliated Hospital of Soochow University; Nana Ping, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No